CLINICAL TRIAL: NCT01600794
Title: To Evaluate The Androgens and Ovary Function Impact on The Pregnancy Outcome in In Vitro Fertilization
Brief Title: To Evaluate The Anrogens and Ovary Function in In Vitro Fertilization
Status: Suspended | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-TMU-IVF-201107012
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: In Vitro Fertilization
Keywords: In Vitro Fertilization (IVF); androgens; ovary function; This study include the patients who are evaluated by the doctors and are sure to process the In Vitro Fertilization cycle.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- male/female, immunity or others factor infertility, IVF

SUMMARY:
Because the society convention is changed, people are late for getting married, leading to increasing the bearing age in women. According to the previous study, if the age is over 30, the oocyte number in ovary has left only 10％ and 3％ in over 40 years old. The data is collected by Bureau of Health Promotion, Department of Health shows that there are about 7000 people treating the infertility and it spends about 150000 to 250000 NT dollars in every in vitro fertilization (IVF) cycle, but the live birth rate is only 30％. So it is important to know how to estimate and approve the ovary function that lead to increase the live birth rate. The investigators plan to estimate the correlation between the serum androgens levels and pregnancy outcome in the women who have infertility problem. Furthermore, for the repeated IVF cycle, the ovary function might be re-evlauated because of the possible effect from stimulated drugs used on previous cycle. It's important to understand the ovary function for IVF patient to choose the appropriate drugs and dose.

The investigators use blood and clinical test to analyze, the items for analysis are below:

1. Routine blood test: FSH、LH、E2、P4、Anti-Mullerian Hormone(AMH)、
2. Studied blood test: Inhibin B、total testosterone (TT)、Androstenedione、DHEA-S
3. Clinical test: Ultrasound
4. Personal condition. In order to finishing the test, every patient will be asked to collect about 10 to 15 cc blood for the research.

ELIGIBILITY:
Inclusion Criteria:

* This study include the patients who are evaluated by the doctors and are sure to process the IVF cycle.

Exclusion Criteria:

* This study exclude the patients who are not evaluated by the doctors and are not sure to process the IVF cycle.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study include the patients who are evaluated by the doctors and are sure to process the IVF cycle.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-10; Study Completion 2012-10 (Estimated)